### **INFORMED CONSENT STATEMENT**

### PARTICIPANT IN MEDICAL RESEARCH BY NANO HYDROGEN BUBBLE INFUSION METHODS





### With Research Title:

# Intravenous hydrogen nanobubbles effect on cardiac physiology and quality of life: a single blind, dose-response study

Malang, Indonesia
19th September, 2022





## INFORMED CONSENT STATEMENT CLINICAL TRIAL PARTICIPANT CONSENT FORM METHOD: INTRAVENOUS HYDROGEN NANOBUBBLE INFUSION

I, the undersigned,

Name :
National ID Number (NIK):
Date of Birth :
Address :
Phone Number :

#### Hereby declare with full awareness that:

- 1. I voluntarily agree to participate as a subject in a medical research study using intravenous hydrogen nanobubble infusion conducted by the Institut Molekul Indonesia, located at Jl. Ciliwung 20–22, Malang, and handled by qualified medical personnel licensed in their respective fields.
- 2. I consent to the use of my personal and medical data as a research subject for the purposes of scientific investigation by Institut Molekul Indonesia.
- 3. After receiving a clear explanation regarding the research method involving intravenous hydrogen nanobubble infusion, I understand, acknowledge, and accept the medical procedure along with any associated risks.
  - 3.1 This research involves intravenous infusion/injection of hydrogen nanobubbles to human subjects in order to improve cardiovascular function and overall quality of life.
  - 3.2 The infusion procedure is administered in stages based on observation and recommendation by the medical team, following these program types:
    - Type A (1st & 2nd infusions)
    - Type B (3rd & 4th infusions)
    - Type C (5th & 6th infusions)
    - Type D (7th & 8th infusions)
    - Type E (9th & 10th infusions)
    - Type F (11th & 12th infusions)
  - 3.3 Following the completion of Types A through F, there may be a follow-up exit program and/or maintenance program if deemed necessary by the clinical team.
- 4. If any medical complications arise as a result of the intervention, I agree to undergo appropriate treatment and recovery procedures under the supervision of the qualified doctors from Institut Molekul Indonesia.





5. Any disputes or outcomes related to this procedure shall be resolved through mutual deliberation and agreement, without resorting to legal action, either criminal or civil.

This statement is made truthfully and voluntarily, with full awareness and without coercion from any party.

| Malang, 19th September, 2022 |
|------------------------------|
| Participant Signature: |
| Witness I: |
| Witness II: |